CLINICAL TRIAL: NCT00834106
Title: A Randomized, Placebo-Controlled, Double-Blind Study of Quadrivalent HPV (Types 6, 11, 16, 18) L1 Virus-Like Particle (VLP) Vaccine to Investigate the Safety, and Efficacy in Chinese 20 - to 45-Years-Old Women
Brief Title: Prevention of Human Papillomavirus (HPV) in 20 to 45 Year Old Chinese Women (V501-041)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V501-041; 2009_532
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2017-10-12 (Actual); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: HPV Infections
Keywords: HPV 6/11/16/18 Infection
MeSH Terms: conditions — Papillomavirus Infections | interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- qHPV (Experimental): Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine administered by intramuscular injection on Day 1, Month 2, and Month 6
  Interventions: Biological: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine
- Placebo (Placebo Comparator): Placebo administered by intramuscular injection on Day 1, Month 2, and Month 6
  Interventions: Biological: Comparator: placebo (unspecified)

INTERVENTIONS:
Biological: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine — Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine injection at Day 1, Month 2, and Month 6.
  Other Names: Gardasil ™; V501
  Arms: qHPV
Biological: Comparator: placebo (unspecified) — Aluminum-containing Vaccine placebo injection at Day 1, Month 2, and Month 6.
  Arms: Placebo

SUMMARY:
A study to test the safety and effectiveness of Quadrivalent HPV (types 6, 11, 16, 18) L1 VLP vaccine against combined incidence of HPV 6/11/16/18-related persistent infection and vaccine type-specific genital disease among Chinese females between the ages of 20 and 45.

DETAILED DESCRIPTION:
The Base Study V501-041 duration was 30 months. The study was extended to further evaluate the efficacy of Quadrivalent HPV (Type 6, 11, 16, 18) L1 VLP (qHPV) vaccine against Cervical Intraepithelial Neoplasia Grade 2 (CIN 2), CIN 3, Adenocarcinoma In Situ (AIS), and/or cervical cancer. The efficacy was followed through the Month 78 visit, and the close-out visit was conducted at approximately Month 90 with only safety data collected

ELIGIBILITY:
Inclusion Criteria:

* Healthy women between the ages of 20 and 45
* Have used effective contraception for 2 weeks prior to starting in the study
* Does not have a temperature within 24 hours before the first injection

Exclusion Criteria:

* Prior history of genital warts
* More than 4 lifetime sexual partners
* Have undergone hysterectomy
* Have active cervical disease or history of cervical disease

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3006 (Actual)
Dates: Start 2008-12-31 (Actual); Primary Completion 2012-05-11 (Actual); Study Completion 2016-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Background] Wei L, Xie X, Liu J, Zhao Y, Chen W, Zhao C, Wang S, Liao X, Shou Q, Qiu Y, Qiao Y, Saah AJ. Efficacy of quadrivalent human papillomavirus vaccine against persistent infection and genital disease in Chinese women: A randomized, placebo-controlled trial with 78-month follow-up. Vaccine. 2019 Jun 12;37(27):3617-3624. doi: 10.1016/j.vaccine.2018.08.009. Epub 2018 Aug 16. PMID 30122646
- [Derived] Chen W, Zhao Y, Xie X, Liu J, Li J, Zhao C, Wang S, Liao X, Shou Q, Zheng M, Saah AJ, Wei L, Qiao Y. Safety of a quadrivalent human papillomavirus vaccine in a Phase 3, randomized, double-blind, placebo-controlled clinical trial among Chinese women during 90 months of follow-up. Vaccine. 2019 Feb 4;37(6):889-897. doi: 10.1016/j.vaccine.2018.12.030. Epub 2019 Jan 9. PMID 30638797

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were stratified by age before randomization: 20 to 26 years of age and 27 to 45 years of age.
Period: Base Study (Day 1 to Month 30)
Arm/Group | qHPV | Placebo
Started | 1503 (Randomized participants) | 1503 (Randomized participants)
Vaccinated | 1503 | 1503
Completed Vaccinations | 1473 | 1463
Completed | 1401 (Completed Month 30 follow-up) | 1358 (Completed Month 30 follow-up)
Not Completed | 102 | 145
Period: Extension Study (Month 42 to Month 90)
Arm/Group | qHPV | Placebo
Started | 1404 (Some participants missed the Month 30 visit but returned for the Month 42 visit) | 1368 (Some participants missed the Month 30 visit but returned for the Month 42 visit)
Completed | 1308 | 1294
Not Completed | 96 | 74

BASELINE CHARACTERISTICS:
Population: All randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | qHPV | Placebo | Total
Number analyzed (Participants) | 1503 | 1503 | 3006
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.7 (6.4) | 28.7 (6.4) | 28.7 (6.4)
Age, Customized [Number; unit: Participants]
  20 to 26 years of age | 923 | 917 | 1840
  27 to 45 years of age | 580 | 586 | 1166
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1503 | 1503 | 3006
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1503 | 1503 | 3006

OUTCOME MEASURES:

1. Primary Outcome: Base Study: Combined Incidence of 6-Month Persistent Infection, Cervical Intraepithelial Neoplasia (CIN+), and External Genital Lesions Related to Human Papillomavirus (HPV) Type 6, 11, 16, or 18 in 20 to 45 Year Old Participants (Test of Hypothesis)
Description: The endpoint included pathology panel consensus diagnosis of 6-month persistent infection, CIN+ (including CIN grade 1, 2, or 3, cervical adenocarcinoma in situ (AIS), and cervical cancer), or external genital lesions related to HPV Types 6, 11, 16, or 18 detected by polymerase chain reaction (PCR) in an adjacent section from the same tissue block.
Time Frame: From Day 1 until >=25 cases accumulate, up to Month 30
Population: The population analyzed included participants who received the full vaccination series, had at least 1 visit after Month 7, had no general protocol violations, and were seronegative at Baseline and polymerase chain reaction-negative from Baseline through Month 7 for HPV types 6, 11, 16, and 18.
Measure: Number; unit: Cases per 100 person-years of follow-up
Units Other Than Participants: person-years
Arm/Group | qHPV | Placebo
Number analyzed (Participants) | 1281 | 1249
Number analyzed (person-years) | 2491 | 2389
Cases per 100 person-years of follow-up | 0.3 | 1.2
Statistical Analysis 1: Comparison: qHPV vs Placebo; Test type: Superiority or Other; Vaccine efficacy = 76.0, 95% CI 2-sided [43.7 to 91.1] — Vaccine efficacy = 100 * [1 - (incidence rate with V501 / incidence rate with placebo)]. The pre-specified success criterion was that the lower bound of the 95% confidence interval for vaccine efficacy excludes 0%

2. Primary Outcome: Base Study: Combined Incidence of 6-Month Persistent Infection, CIN+, and External Genital Lesions Related to Human Papillomavirus (HPV) Type 6, 11, 16, or 18 in 20 to 26 Years Old Participants (Test of Hypothesis)
Description: The endpoint included pathology panel consensus diagnosis of 6-month persistent infection, CIN+ (including CIN grade 1, 2, or 3, cervical adenocarcinoma in situ (AIS), and cervical cancer), or external genital lesions related to HPV Types 6, 11, 16, or 18 detected by PCR in an adjacent section from the same tissue block.
Time Frame: From Day 1 until >=17 cases accumulate, up to Month 30
Population: The population analyzed included participants 20 to 26 years old at Baseline who received the full vaccination series, had at least 1 visit after Month 7, had no general protocol violations, and were seronegative at Baseline and polymerase chain reaction-negative from Baseline through Month 7 for HPV types 6, 11, 16, and 18.
Measure: Number; unit: Cases per 100 person-years of follow-up
Units Other Than Participants: person-years
Arm/Group | qHPV | Placebo
Number analyzed (Participants) | 760 | 733
Number analyzed (person-years) | 1461 | 1376
Cases per 100 person-years of follow-up | 0.2 | 1.2
Statistical Analysis 1: Comparison: qHPV vs Placebo; Test type: Superiority or Other; Vaccine efficacy = 82.3, 95% CI 2-sided [38.3 to 96.7] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Entire Study: Combined Incidence of CIN2+ Related to HPV Types 16 or 18 in 20 to 45 Year Old Participants (End of Study Test of Hypothesis)
Description: The endpoint included pathology panel consensus diagnosis of CIN2+ (including CIN grade 2 or 3, AIS, and cervical cancer) related to HPV Types 16 or 18 detected by PCR in an adjacent section from the same tissue block.
Time Frame: Up to Month 78
Population: The population analyzed included participants who received the full vaccination series, had at least 1 visit after Month 7, had no general protocol violations, and were seronegative at Baseline and polymerase chain reaction-negative from Baseline through Month 7 for HPV types 16 and 18.
Measure: Number; unit: Cases per 100 person-years of follow-up
Units Other Than Participants: person-years
Arm/Group | qHPV | Placebo
Number analyzed (Participants) | 1265 | 1237
Number analyzed (person-years) | 6992 | 6789
Cases per 100 person-years of follow-up | 0.0 | 0.1
Statistical Analysis 1: Comparison: qHPV vs Placebo; Test type: Superiority or Other; p = 0.0072, Exact test, 1-sided; Vaccine efficacy = 100, 95% CI 2-sided [32.3 to 100] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Base Study: Percentage of Participants With One or More Solicited Injection-site Adverse Events
Description: An adverse event (AE) is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the sponsor's product, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the sponsor's product, is also an AE. Injection-site AEs were prompted on the Vaccination Report Card (VRC), which was completed by the participant for 15 days after each vaccination.
Time Frame: Up to 15 days after any vaccination
Population: All vaccinated participants with safety follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | qHPV | Placebo
Number analyzed (Participants) | 1499 | 1498
Percentage of participants | 37.6 | 27.8

5. Primary Outcome: Base Study: Percentage of Participants With One or More Systemic Adverse Events
Description: An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the sponsor's product, whether or not considered related to the use of the product. Any worsening of a preexisting condition which is temporally associated with the use of the sponsor's product, is also an AE.
Time Frame: Up to 15 days after any vaccination
Population: All vaccinated participants with safety follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | qHPV | Placebo
Number analyzed (Participants) | 1499 | 1498
Percentage of participants | 50.4 | 48.7

6. Primary Outcome: Base Study: Percentage of Participants Discontinued From Study Vaccination Due to an Adverse Event
Description: as for outcome 5
Time Frame: Up to 6 months
Population: All vaccinated participants with safety follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | qHPV | Placebo
Number analyzed (Participants) | 1499 | 1498
Percentage of participants | 0.1 | 0.2

7. Primary Outcome: Entire Study: Percentage of Participants With One or More Vaccine-related Serious Adverse Events
Description: A serious adverse event (SAE) is an AE that results in death, is life threatening, results in persistent or significant disability or incapacity, results in or prolongs a hospitalization, is a congenital anomaly or birth defect, is an overdose or, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention. Related SAEs were those deemed possibly, probably, or definitely related to study vaccine or a study procedure.
Time Frame: Up to approximately 90 months
Population: All vaccinated participants with safety follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | qHPV | Placebo
Number analyzed (Participants) | 1499 | 1498
Percentage of participants | 0.0 | 0.1

8. Primary Outcome: Entire Study: Percentage of Participants Who Died
Description: The percentage of participants who died on study due to any cause, whether or not related to the investigational product, were reported for each arm
Time Frame: Up to approximately 90 months
Population: All vaccinated participants with safety follow-up
Measure: Number; unit: Percentage of participants
Arm/Group | qHPV | Placebo
Number analyzed (Participants) | 1499 | 1498
Percentage of participants | 0.1 | 0.0

9. Secondary Outcome: Entire Study: Combined Incidence of 12-Month Persistent Infection, CIN+, and External Genital Lesions Related to Human Papillomavirus (HPV) Type 6, 11, 16, or 18 in 20 to 45 Year Old Participants (End of Study Update)
Description: The endpoint included pathology panel consensus diagnosis of 12-month persistent infection, CIN+ (including CIN grade 1, 2, or 3, cervical adenocarcinoma in situ (AIS), and cervical cancer), or external genital lesions related to HPV Types 6, 11, 16, or 18 detected by PCR in an adjacent section from the same tissue block.
Time Frame: Up to 78 months
Population: as for outcome 1
Measure: Number; unit: Cases per 100 person-years of follow-up
Units Other Than Participants: person-years
Arm/Group | qHPV | Placebo
Number analyzed (Participants) | 1281 | 1249
Number analyzed (person-years) | 8515 | 8015
Cases per 100 person-years of follow-up | 0.1 | 0.7
Statistical Analysis 1: Comparison: qHPV vs Placebo; Test type: Superiority or Other; Vaccine efficacy = 91.8, 95% CI 2-sided [79.8 to 97.4] — Vaccine efficacy = 100 * [1 - (incidence rate with V501 / incidence rate with placebo)]

10. Secondary Outcome: Entire Study: Combined Incidence of 12-Month Persistent Infection, CIN+, and External Genital Lesions Related to Human Papillomavirus (HPV) Type 6, 11, 16, or 18 in 20 to 26 Year Old Participants (End of Study Update)
Description: as for outcome 9
Time Frame: Up to 78 months
Population: The population analyzed included participants 20 to 26 years of age at Baseline who received the full vaccination series, had at least 1 visit after Month 7, had no general protocol violations, and were seronegative at Baseline and polymerase chain reaction-negative from Baseline through Month 7 for HPV types 6, 11, 16, and 18.
Measure: Number; unit: Cases per 100 person-years of follow-up
Units Other Than Participants: person-years
Arm/Group | qHPV | Placebo
Number analyzed (Participants) | 760 | 733
Number analyzed (person-years) | 4952 | 4559
Cases per 100 person-years of follow-up | 0.0 | 0.6
Statistical Analysis 1: Comparison: qHPV vs Placebo; Test type: Superiority or Other; Vaccine efficacy = 93.2, 95% CI 2-sided [72.9 to 99.2] — Vaccine efficacy = 100 * [1 - (incidence rate with V501 / incidence rate with placebo)]

ADVERSE EVENTS:
Time Frame: Up to approximately 90 months
Description: All vaccinated participants with safety follow-up
Arm/Group | qHPV | Placebo
Serious Adverse Events (participants affected / at risk) | 38/1499 | 43/1498
Other Adverse Events (participants affected / at risk) | 876/1499 | 799/1498
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | qHPV (N=1499) | Placebo (N=1498)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Thyroid Mass (Endocrine disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Meniscus Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Benign Hydatidiform Mole (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fibroadenoma Of Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intraductal Papilloma Of Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian Cancer Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian Germ Cell Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Phyllodes Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 7 (7)
Vaginal Cancer Stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carpal Tunnel Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular Disorder (Nervous system disorders) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Trigeminal Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Abortion Missed (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Cephalo-Pelvic Disproportion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 3 (3)
Foetal Damage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Foetal Death (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Gestational Hypertension (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 0 (0)
Placenta Accreta (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral Cyst (Renal and urinary disorders) | 1 (1) | 0 (0)
Cervical Dysplasia (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Cervical Polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Endometrial Hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Fallopian Tube Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic Fluid Collection (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine Disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine Polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Epiglottic Cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Appendicectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Ectopic Pregnancy Termination (Surgical and medical procedures) | 0 (0) | 1 (1)
Fallopian Tube Operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Haemorrhoid Operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Labour Induction (Surgical and medical procedures) | 0 (0) | 1 (1)
Myomectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Synovial Cyst Removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Thyroid Adenoma Removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Thyroid Nodule Removal (Surgical and medical procedures) | 1 (1) | 1 (1)
Uterine Polypectomy (Surgical and medical procedures) | 3 (4) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | qHPV (N=1499) | Placebo (N=1498)
Diarrhoea (Gastrointestinal disorders) | 89 (106) | 94 (105)
Nausea (Gastrointestinal disorders) | 100 (122) | 95 (106)
Fatigue (General disorders) | 227 (310) | 193 (247)
Injection Site Erythema (General disorders) | 176 (233) | 133 (163)
Injection Site Induration (General disorders) | 115 (151) | 64 (76)
Injection Site Pain (General disorders) | 494 (778) | 346 (450)
Injection Site Pruritus (General disorders) | 113 (145) | 77 (83)
Injection Site Swelling (General disorders) | 160 (220) | 78 (92)
Pyrexia (General disorders) | 388 (493) | 352 (432)
Myalgia (Musculoskeletal and connective tissue disorders) | 224 (307) | 153 (185)
Headache (Nervous system disorders) | 218 (274) | 193 (240)
Cough (Respiratory, thoracic and mediastinal disorders) | 84 (103) | 91 (99)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission.